CLINICAL TRIAL: NCT05015478
Title: Phase 1 - The Use of Rhythmic Light Therapy to Entrain Gamma Oscillations and the Circadian System in Patients With Alzheimer's Disease
Brief Title: Rhythmic Light Therapy for Alzheimer's Disease Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Mariana Figueiro, Professor, Population Health Science and Policy, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: GCO 21-0378-01; 5R01AG072762 (NIH)
Record Dates: First submitted 2021-08-12; First posted 2021-08-20 (Actual); Results first posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Mild Cognitive Impairment
Keywords: Light Treatment; Circadian Rhythms; Gamma Wave Entrainment; Rhythmic Light; Mild Alzheimer's Disease; Sleep; Memory; Electroencephalogram
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Tailored Rhythmic Lighting then Inactive Placebo Rhythmic Lighting (Active Comparator): 1. hour intervention period where active lighting is experienced by participants. then 1 hour intervention period where an inactive, placebo lighting condition is experienced by participants.
  2. sessions, 1 week apart
  Interventions: Device: Tailored Rhythmic Lighting Intervention
- Inactive Placebo Rhythmic Lighting then Active Tailored Rhythmic Lighting (Placebo Comparator): 1. hour intervention period where an inactive, placebo lighting condition is experienced by participants. then 1 hour intervention period where active lighting is experienced by participants.
  2. sessions, 1 week apart
  Interventions: Device: Placebo Rhythmic Lighting Intervention

INTERVENTIONS:
Device: Tailored Rhythmic Lighting Intervention — 40 hertz (Hz) rhythmic lighting (RL) for a duration of 1 hour. The flicker frequency of the 40 Hz RL will be 40 Hz and the stimulation will be a square wave with a 50 % duty cycle (i.e., 12.5 milliseconds light- on and 12.5 milliseconds light-off). The RL will provide a 30 lux of red light on a vertical plane at the eye level.
  Arms: Active Tailored Rhythmic Lighting then Inactive Placebo Rhythmic Lighting
Device: Placebo Rhythmic Lighting Intervention — Placebo rhythmic light (RL) for a duration of 1 hour. In the placebo RL condition, the duty cycle will be delivered at randomly varying frequencies of 20 Hz and 50 Hz, specifically avoiding the frequency of 40 Hz. The placebo RL conditions will provide a 30 lux of red light on a vertical plane at the eye level.
  Arms: Inactive Placebo Rhythmic Lighting then Active Tailored Rhythmic Lighting

SUMMARY:
The investigator will investigate how light delivering 40 hertz (Hz) affects subjective sleep and cognition in a controlled laboratory study. A lab study will allow the collection of electroencephalogram (EEG) data, perform cognitive tests, and observe the response in those with mild cognitive impairment (MCI) compared to a healthy control group (HC).

Participants will attend two study sessions over the course of two weeks. During both sessions, all participants will experience 10 minutes of a low-level light, followed by a data collection period which involves a sleepiness rating, an electroencephalogram (EEG) recording, and a computerized memory test. Participants will then experience either a RL or a placebo RL condition for one hour, after which there will be a second data collection.

DETAILED DESCRIPTION:
The investigator will demonstrate the effect of 40 hertz (Hz) rhythmic light (RL) to promote gamma wave entrainment (rhythmic light [RL]) on: brain response (electroencephalography [EEG]); cognitive performance (working memory task); and subjective sleepiness (questionnaires). The study will recruit 20 adult mild cognitive impairment (MCI) patients and 20 healthy, age-matched controls (HC) to participate in this study.

Sessions will initiate with a 10-minute adaptation period to a low-level ambient light providing illuminance of 15 lux at participants' eye level on a vertical plane, followed by a pre-exposure data collection period, including Karolinska Sleepiness Scale (KSS), EEG, and a working memory task. Participants will experience either 40 Hz RL or placebo RL conditions for a duration of 1 hour, followed by the second data collection period. On the second data collection day, participants will experience the other condition, so that all participants experience both lighting conditions. The experimental sessions will start at 14:00 on each experimental day which will be separated by 1 week.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be diagnosed with amnestic mild cognitive impairment or mild Alzheimer's disease, as defined by a Montreal Cognitive Assessment (MoCA) score between 17 and 25
* For the age-matched healthy controls, participants must not be diagnosed with mild cognitive impairment or Alzheimer's disease related dementias (MoCA score above 25).
* Participants must score a 5 or less in the Pittsburgh Sleep Quality Index (PSQI)

Exclusion Criteria:

* All participants must not be taking sleeping medication or oral melatonin
* Presence of another brain disease that fully explains the dementia (extensive brain vascular disease, Parkinson's disease, dementia with Lewy bodies, traumatic brain injury, or multiple sclerosis)
* residence in a skilled nursing facility or long-term care
* Major organ failure (e.g., kidney failure)
* Uncontrolled generalized disorders such as hypertension or diabetes
* Obstructing cataracts, macular degeneration, and blindness
* Severe sleep apnea or restless leg syndrome
* History of epilepsy

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2023-07-12 (Actual); Study Completion 2023-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mariana Figueiro, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (2):
- United States (2):
  - Light and Health Research Center, Menands, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York

REFERENCES:
- [Background] Akerstedt T, Gillberg M. Subjective and objective sleepiness in the active individual. Int J Neurosci. 1990 May;52(1-2):29-37. doi: 10.3109/00207459008994241. PMID 2265922
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Hoch CC, Yeager AL, Kupfer DJ. Quantification of subjective sleep quality in healthy elderly men and women using the Pittsburgh Sleep Quality Index (PSQI). Sleep. 1991 Aug;14(4):331-8. PMID 1947597

RESULTS

PARTICIPANT FLOW:
Groups:
- Health Control Group 1: Healthy Control - Active Tailored Rhythmic Lighting then Inactive Placebo Rhythmic Lighting
  1 hour intervention period where active lighting is experienced by participants. then 1 hour intervention period where an inactive, placebo lighting condition is experienced by participants.
- Health Control Group 2: Healthy Control - Inactive Placebo Rhythmic Lighting then Active Tailored Rhythmic Lighting
  1 hour intervention period where an inactive, placebo lighting condition is experienced by participants. then 1 hour intervention period where active lighting is experienced by participants.
- Mild Cognitive Impairment Group 1: Mild Cognitive Impairment - Active Tailored Rhythmic Lighting then Inactive Placebo Rhythmic Lighting
  1 hour intervention period where active lighting is experienced by participants. then 1 hour intervention period where an inactive, placebo lighting condition is experienced by participants.
- Mild Cognitive Impairment Group 2: Mild Cognitive Impairment - Inactive Placebo Rhythmic Lighting then Active Tailored Rhythmic Lighting
  1 hour intervention period where an inactive, placebo lighting condition is experienced by participants. then 1 hour intervention period where active lighting is experienced by participants.
Period: Initial Experimental Condition
Arm/Group | Health Control Group 1 | Health Control Group 2 | Mild Cognitive Impairment Group 1 | Mild Cognitive Impairment Group 2
Started | 11 | 15 | 12 | 14
Completed | 11 | 15 | 12 | 14
Not Completed | 0 | 0 | 0 | 0
Period: Second Experimental Condition
Arm/Group | Health Control Group 1 | Health Control Group 2 | Mild Cognitive Impairment Group 1 | Mild Cognitive Impairment Group 2
Started | 11 | 15 | 12 | 14
Completed | 11 | 15 | 12 | 13
Not Completed | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Health Control: Health Participants - 1 hour intervention period where active lighting is experienced by participants or 1 hour intervention period where an inactive, placebo lighting condition is experienced by participants then in the second intervention experiences the opposite of the first intervention.
- Mild Cognitive Impairment: Participants with Mild Cognitive Impairment - 1 hour intervention period where active lighting is experienced by participants or 1 hour intervention period where an inactive, placebo lighting condition is experienced by participants then in the second intervention experiences the opposite of the first intervention.
- Total: Total of all reporting groups
Arm/Group | Health Control | Mild Cognitive Impairment | Total
Number analyzed (Participants) | 26 | 26 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 16 | 16 | 32
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 32
  Male | 10 | 10 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 21 | 21 | 42
  Unknown or Not Reported | 4 | 4 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 19 | 19 | 38
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Electroencephalography (EEG) Power at 40 Hertz (Hz)
Description: Electroencephalography (EEG) recordings - the change in 40 Hz gamma power, computed by calculating the difference between the average gamma power at baseline (T1) and during the light intervention (T2). This difference was obtained by subtracting baseline 40 Hz power from the intervention 40 Hz power to assess acute neural effects
Time Frame: baseline and during the light intervention
Population: EEG data not collected for first 12 participants. Protocol revised to include EEG data collection subsequently.
Measure: Mean (Standard Deviation); unit: μV2/Hz
Groups:
- MCI - Inactive Placebo Rhythmic Lighting; HC - Placebo Rhythmic Lighting: 1 hour intervention period where an inactive, placebo lighting condition is experienced by participants.
  Placebo Rhythmic Lighting Intervention: Placebo rhythmic light (RL) for a duration of 1 hour. In the placebo RL condition, the duty cycle will be delivered with a random interval determined by a Poisson process with an average interval of 40 hertz (Hz). The placebo RL conditions will provide a 30 lux of red light on a vertical plane at the eye level.
- MCI - Active Tailored Rhythmic Lighting; HC - Active Tailored Rhythmic Lighting: 1 hour intervention period where active lighting is experienced by participants.
  Tailored Rhythmic Lighting Intervention: 40 hertz (Hz) rhythmic lighting (RL) for a duration of 1 hour. The flicker frequency of the 40 Hz RL will be 40 Hz and the stimulation will be a square wave with a 50 % duty cycle (i.e., 12.5 milliseconds light- on and 12.5 milliseconds light-off). The RL will provide a 30 lux of red light on a vertical plane at the eye level.
Arm/Group | MCI - Inactive Placebo Rhythmic Lighting | MCI - Active Tailored Rhythmic Lighting | HC - Placebo Rhythmic Lighting | HC - Active Tailored Rhythmic Lighting
Number analyzed (Participants) | 10 | 10 | 10 | 10
μV2/Hz
  Oz | 3.54 (0.43) | 5.28 (0.82) | 2.83 (0.53) | 4.10 (0.66)
  Pz | 2.69 (0.53) | 5.24 (0.94) | 3.86 (0.51) | 3.56 (0.55)
  POz | 2.87 (0.43) | 5.18 (0.88) | 3.29 (0.51) | 3.57 (0.64)

2. Secondary Outcome: Mean Change in Subjective Sleepiness Using the Karolinska Sleepiness Scale (KSS)
Description: The Karolinska Sleepiness Scale (KSS) outcome prompts participants to rate how sleepy or alert they are feeling on a scale ranging from 1 to 9, where 1 = "very alert," 3 = "rather alert," 5 = "neither alert nor sleepy," 7 = "sleepy, but no difficulty remaining awake," and 9 = "very sleepy, fighting sleep, an effort to remain awake."
Time Frame: Baseline and 1 hour after intervention (intervention is 2 hours)
Population: EEG data not collected for first 12 participants. Protocol revised to include EEG data collection subsequently.
  Outcome measure is comparing the two interventions Active Tailored Rhythmic Lighting vs Inactive Placebo Rhythmic Lighting regardless of cognitive status.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Active Tailored Rhythmic Lighting: 1 hour intervention period where active lighting is experienced by participants.
  Tailored Rhythmic Lighting Intervention: 40 hertz (Hz) rhythmic lighting (RL) for a duration of 1 hour. The flicker frequency of the 40 Hz RL will be 40 Hz and the stimulation will be a square wave with a 50 % duty cycle (i.e., 12.5 milliseconds light- on and 12.5 milliseconds light-off). The RL will provide a 30 lux of red light on a vertical plane at the eye level.
- Inactive Placebo Rhythmic Lighting: 1 hour intervention period where an inactive, placebo lighting condition is experienced by participants.
  Placebo Rhythmic Lighting Intervention: Placebo rhythmic light (RL) for a duration of 1 hour. In the placebo RL condition, the duty cycle will be delivered with a random interval determined by a Poisson process with an average interval of 40 hertz (Hz). The placebo RL conditions will provide a 30 lux of red light on a vertical plane at the eye level.
Arm/Group | Active Tailored Rhythmic Lighting | Inactive Placebo Rhythmic Lighting
Number analyzed (Participants) | 40 | 40
score on a scale | 0.44 (0) | 0.49 (0)

3. Secondary Outcome: Cognition Using a Working Memory Task
Description: Participants view a serial visual display of letters and math problems. They are asked to hold the letters in memory while simultaneously determining if the simple math problems are correct (e.g., 7+5=13). Performance is assessed in percent correct and by measuring accuracy and Reaction Time (RT).
Time Frame: 1 hour after intervention (intervention is 2 hours)
Reporting Status: Not Posted, anticipated posting 2025-12

ADVERSE EVENTS:
Time Frame: 2 hours
Groups:
- MCI - Inactive Placebo Rhythmic Lighting; HC - Active Tailored Rhythmic Lighting; MC - Inactive Placebo Rhythmic Lighting: 1 hour intervention period where active lighting is experienced by participants.
  Tailored Rhythmic Lighting Intervention: 40 hertz (Hz) rhythmic lighting (RL) for a duration of 1 hour. The flicker frequency of the 40 Hz RL will be 40 Hz and the stimulation will be a square wave with a 50 % duty cycle (i.e., 12.5 milliseconds light- on and 12.5 milliseconds light-off). The RL will provide a 30 lux of red light on a vertical plane at the eye level.
Arm/Group | MCI - Active Tailored Rhythmic Lighting | MCI - Inactive Placebo Rhythmic Lighting | HC - Active Tailored Rhythmic Lighting | MC - Inactive Placebo Rhythmic Lighting
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/26 | 0/26 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26 | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 0/26 | 0/26 | 0/26 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-02-01): https://cdn.clinicaltrials.gov/large-docs/78/NCT05015478/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-01): https://cdn.clinicaltrials.gov/large-docs/78/NCT05015478/SAP_001.pdf